CLINICAL TRIAL: NCT00584584
Title: A Proof of Concept Study of the Effects of QAX576 (an Interleukin-13 Monoclonal Antibody) on Allergic Inflammation Following Out of Allergy Season Repeated Nasal Allergen Challenge in Subjects With Seasonal Allergic Rhinitis Sensitive to Timothy Grass Pollen
Brief Title: An Exploratory Study of the Effects of a Single Dose of QAX576 (an Interleukin-13 Monoclonal Antibody) on Simulated Hayfever
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQAX576A2104
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Allergic Rhinitis
Keywords: Allergic rhinitis, adults, monoclonal antibody, interleukin-13.
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: QAX576
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QAX576
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
This study will investigate whether a single dose QAX576 (an interleukin-13 monoclonal antibody) gives protection against a model of hayfever

ELIGIBILITY:
Inclusion Criteria:

* History of allergic rhinitis.

Exclusion Criteria:

* Respiratory disease other than mild intermittent asthma.
* Received immunotherapy in past 3 years.
* History of clinically significant drug allergy.
* History of clinical schistosomiasis or travel within 6 months prior to or following study to an area with endemic schistosomiasis.
* History of exposure to human therapeutic antibodies, immunoglobulins or other plasma products.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-12; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Markers of allergic inflammation in the nose measured over 5-8 days post-dose. | throughout the study

SECONDARY OUTCOMES:
- Nasal symptom scores over 5-8 days post-dose. - Blood levels of QAX576 to 3 months post-dose. - Marker of allergic inflammation in blood to 3 months post-dose. | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: NOVARTIS, Principal Investigator — Novartis investigator site
Locations (2):
- Novartis Investigator Site, Hanover, Germany
- Novartis Investigator Site, London, United Kingdom

REFERENCES:
- See also: Results of CQAX576A2104 from United European Gastroenterology journal — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4212306/